CLINICAL TRIAL: NCT06657833
Title: DEBSCAN-IVL. Drug Eluting Balloon or Drug Eluting Stent to Treat CAlcified Nodules After IntraVascular Lithotripsy.
Acronym: DEBSCAN-IVL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación EPIC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EPIC40-DEBSCAN-IVL
Record Dates: First submitted 2024-10-21; First posted 2024-10-26 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Coronary Artery Disease
Keywords: Calcified Nodules; Calcified lesions; Drug eluting balloon; Drug eluting stent
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drug Eluting Balloon (DEB) (Other)
  Interventions: Device: Percutaneous coronary intervention of a calcified nodule with intravascular lithotripsy followed by drug eluting balloon
- Drug Eluting Stent (DES) (Other)
  Interventions: Device: Percutaneous coronary intervention of a calcified nodule with intravascular lithotripsy followed by drug eluting stent

INTERVENTIONS:
Device: Percutaneous coronary intervention of a calcified nodule with intravascular lithotripsy followed by drug eluting balloon — Percutaneous coronary intervention of a calcified nodule with intravascular lithotripsy followed by drug eluting balloon
  Arms: Drug Eluting Balloon (DEB)
Device: Percutaneous coronary intervention of a calcified nodule with intravascular lithotripsy followed by drug eluting stent — Percutaneous coronary intervention of a calcified nodule with intravascular lithotripsy followed by drug eluting stent
  Arms: Drug Eluting Stent (DES)

SUMMARY:
International, investigator-driven, multicenter, open-label, prospective randomized controlled trial where patients with de novo lesions due to calcified nodules (CN) were randomized to drug eluting balloon (DEB) or drug eluting stents (DES).

DETAILED DESCRIPTION:
Regardless some observational data of DEB performance in calcified lesions, there is a lack of data about the safety and efficacy in the setting of calcified nodules. However, a "leave-nothing-behind" PCI strategy is attractive in this scenario in which the probability of non-optimal stent expansion and apposition is higher, hypothesis is, that following optimal plaque modification with IVL, the utilization of a DEB is either non-inferior or possibly superior to DES in terms of late lumen loss and net luminal gain at 6 months follow up.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all inclusion criteria:

* Patients >18 years admitted for stable coronary artery disease or acute coronary syndromes and indication for percutaneous coronary intervention (PCI) and
* Severe coronary lesion with calcified nodule, confirmed with intracoronary imaging (optical coherence tomography or intravascular ultrasound) and;
* Lesion to treat in a vessel between 2.5 and 4 mm.

Exclusion Criteria:

Patients must not meet any criteria

* Inability to provide oral and written informed consent or unwillingness to come back for systematic angiographic follow-up.
* Pregnant or breastfeeding patients.
* Cardiogenic Shock or Cardiac arrest at the moment of the index procedure.
* Impossibility to maintain double antiplatelet treatment during at least 1 month.
* Life expectancy <1 year.
* Index lesion at left main stem.
* Aorto-ostial lesion.
* Target lesion previously treated with stents or DEB.
* High thrombus burden in the target lesion (TIMI thrombus scale≥3).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2024-12-17 (Actual); Primary Completion 2027-10-30 (Estimated); Study Completion 2027-10-30 (Estimated)

PRIMARY OUTCOMES:
EFFICACY: Late Lumen Loss (LLL) | 9 Month
  Late lumen loss (LLL, expressed in mm) measured within the treated segment by quantitative coronary angiography (QCA) as the difference between minimal luminal diameter (MLD) at the end of the interventional procedure and MLD at 9-month follow-up
EFFICACY: Net Lumen Gain (NLG) | 9 Month
  Net lumen gain (NLG, expressed in mm) measured by quantitative coronary angiography (QCA) as the difference between minimal luminal diameter within the treated segment (MLD) at 9-month follow-up and MLD at the lesion site at baseline

SECONDARY OUTCOMES:
SAFETY: Dissection | During Percutaneous Coronary Intervention (PCI)
  Freedom from dissection
SAFETY: Perforation | During Percutaneous Coronary Intervention (PCI)
  Freedom from perforation
SAFETY: Abrupt vessel closure | During Percutaneous Coronary Intervention (PCI)
  Freedom from abrupt vessel closure
SAFETY: Slow Flow | During Percutaneous Coronary Intervention (PCI)
  Freedom from slow flow
SAFETY: No Reflow | During Percutaneous Coronary Intervention (PCI)
  Freedom from no reflow
SAFETY: Thrombosis | During Percutaneous Coronary Intervention (PCI)
  Freedom from thrombosis
SAFETY: MACE | Up to 30 days
  Freedom of The composite of cardiac death, myocardial infarction (MI) and target lesion revascularization.
SAFETY: Stent Thrombosis | During hospitalization
  Freedom Stent thrombosis
SAFETY: Major bleeding event | During hospitalization
  Freedom from Mayor bleeding event according to ≥ (BARC 3 criteria )
SAFETY: Stent Thrombosis | During hospitalization
  Freedom from stent thrombosis
SAFETY: Hemodynamic stability | During hospitalization
  Freedom for need for unplanned vasopressors/inotropes or ventricular support devices
EFFICACY: Minimal Lumen Diameter (MLD) | Day 0
  Change in MLD Immediately before procedure, immediately after procedure
EFFICACY: Diameter Stenosis | Day 0
  Percentaje of Diammeter Stenosis after PCI
EFFICACY: Minimal Lumen Diameter (MLD) | 9 Months
  Change in MLD during follow-up
EFFICACY: Minimal Lumen Diammeter (MLD) | 12 Months
  Change in MLD during follow-up
EFFICACY: Binary reestenosis | 9 Months
  Freedom from reestenosis by angiography during follow-up
EFFICACY: Crossover rate | Day 0
  Rate of stent change ( DEB to DES or DES to DEB) during follow-up
SAFETY: MACE | 9 Months
  Freedom of The composite of cardiac death, myocardial infarction (MI) and target lesion revascularization.
SAFETY: MACE | 12 Months
  Freedom of The composite of cardiac death, myocardial infarction (MI) and target lesion revascularization.
SAFETY: MACE | 24 Months
  Freedom of The composite of cardiac death, myocardial infarction (MI) and target lesion revascularization.
SAFETY: Myocardial Infarction | 9 Months
  Freedom from myocardial infarction
SAFETY: Myocardial Infarction | 12 Months
  Freedom from myocardial infarction
SAFETY: Myocardial Infarction | 24 Months
  Freedom from myocardial infarction
SAFETY: Cardiac death | 12 Months
  Freedom from cardiac death
SAFETY: Cardiac death | 24 Months
  Freedom from cardiac death
SAFETY: Target Lesion Revascularization. | 9 Months
  Freedom from TLR
SAFETY: Target Lesion Revascularization. | 12 Months
  Freedom from TLR
SAFETY: Target Lesion Revascularization. | 24 Months
  Freedom from TLR

CONTACTS AND LOCATIONS:
Locations (12):
- Spain (12):
  - Hospital Del Mar, Barcelona
  - Hospital Universitario de La Paz, Fuencarral-El Pardo
  - Hospital Universitario de Galdakao-Usansolo, Galdakao
  - Hospital Universitario de León, León
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Puerta de Hierro, Madrid
  - Hospital Clínico San Carlos, Moncloa-Aravaca
  - Hospital Universitario de Navarra, Pamplona
  - Hospital General Universitario de Valencia, Valencia
  - Hospital Universitario y Politécnico La Fe, Valencia
  - Hospital Clínico Universitario de Valladolid, Valladolid
  - Hospital Universitario de Vigo, Vigo

REFERENCES:
- [Background] Jurado-Román A, Gómez-Menchero A, Gonzalo N, et al. Plaque modification techniques to treat calcified coronary lesions. Position paper from the ACI-SEC. REC Interv Cardiol Engl Ed. Published online February 7, 2023:9672. doi:10.24875/RECICE.M22000345
- [Background] Morofuji T, Kuramitsu S, Shinozaki T, Jinnouchi H, Sonoda S, Domei T, Hyodo M, Shirai S, Ando K. Clinical impact of calcified nodule in patients with heavily calcified lesions requiring rotational atherectomy. Catheter Cardiovasc Interv. 2021 Jan 1;97(1):10-19. doi: 10.1002/ccd.28896. Epub 2020 Apr 7. PMID 32259392
- [Background] Lee T, Mintz GS, Matsumura M, Zhang W, Cao Y, Usui E, Kanaji Y, Murai T, Yonetsu T, Kakuta T, Maehara A. Prevalence, Predictors, and Clinical Presentation of a Calcified Nodule as Assessed by Optical Coherence Tomography. JACC Cardiovasc Imaging. 2017 Aug;10(8):883-891. doi: 10.1016/j.jcmg.2017.05.013. PMID 28797410
- [Background] Sato T, Matsumura M, Yamamoto K, Shlofmitz E, Moses JW, Khalique OK, Thomas SV, Tsoulios A, Cohen DJ, Mintz GS, Shlofmitz RA, Jeremias A, Ali ZA, Maehara A. Impact of Eruptive vs Noneruptive Calcified Nodule Morphology on Acute and Long-Term Outcomes After Stenting. JACC Cardiovasc Interv. 2023 May 8;16(9):1024-1035. doi: 10.1016/j.jcin.2023.03.009. PMID 37164599
- [Background] Ali ZA, Nef H, Escaned J, Werner N, Banning AP, Hill JM, De Bruyne B, Montorfano M, Lefevre T, Stone GW, Crowley A, Matsumura M, Maehara A, Lansky AJ, Fajadet J, Di Mario C. Safety and Effectiveness of Coronary Intravascular Lithotripsy for Treatment of Severely Calcified Coronary Stenoses: The Disrupt CAD II Study. Circ Cardiovasc Interv. 2019 Oct;12(10):e008434. doi: 10.1161/CIRCINTERVENTIONS.119.008434. Epub 2019 Sep 25. PMID 31553205
- [Background] Ho HH, Lee JH, Khoo DZL, Hpone KKS, Li KFC. Shockwave intravascular lithotripsy and drug-coated balloon angioplasty in calcified coronary arteries: preliminary experience in two cases. J Geriatr Cardiol. 2021 Aug 28;18(8):689-691. doi: 10.11909/j.issn.1671-5411.2021.08.009. No abstract available. PMID 34527034
- [Background] Iwasaki Y, Koike J, Ko T, Funatsu A, Kobayashi T, Ikeda T, Nakamura S. Comparison of drug-eluting stents vs. drug-coated balloon after rotational atherectomy for severely calcified lesions of nonsmall vessels. Heart Vessels. 2021 Feb;36(2):189-199. doi: 10.1007/s00380-020-01684-z. Epub 2020 Aug 28. PMID 32857188